CLINICAL TRIAL: NCT05552495
Title: A Phase I Clinical Trial to Evaluate the Tolerability and the Pharmacokinetics of CKD-386 With Co-administration of D013, D326, and D337 in Healthy Adult Volunteers
Brief Title: Clinical Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-386 in Healthy Volunteers Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A83_09BE2219P
Record Dates: First submitted 2022-09-21; First posted 2022-09-23 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Hypertension and Dyslipidemia
MeSH Terms: conditions — Hypertension; Dyslipidemias

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Reference-Test1-Test2 (Experimental)
  Interventions: Drug: CKD-386(4) F1; Drug: CKD-386(4) F2; Drug: D013, D326, D337
- Reference-Test2-Test1 (Experimental)
  Interventions: Drug: CKD-386(4) F1; Drug: CKD-386(4) F2; Drug: D013, D326, D337
- Test1-Reference-Test2 (Experimental)
  Interventions: Drug: CKD-386(4) F1; Drug: CKD-386(4) F2; Drug: D013, D326, D337
- Test1-Test2-Reference (Experimental)
  Interventions: Drug: CKD-386(4) F1; Drug: CKD-386(4) F2; Drug: D013, D326, D337
- Test2-Reference-Test1 (Experimental)
  Interventions: Drug: CKD-386(4) F1; Drug: CKD-386(4) F2; Drug: D013, D326, D337
- Test2-Test1-Reference (Experimental)
  Interventions: Drug: CKD-386(4) F1; Drug: CKD-386(4) F2; Drug: D013, D326, D337

INTERVENTIONS:
Drug: CKD-386(4) F1 — 1 Tablet
  Other Names: Test1
Drug: CKD-386(4) F2 — 1 Tablet
  Other Names: Test2
Drug: D013, D326, D337 — D013 1 Tablet, D326 1Tablet, D337 1 Tablet
  Other Names: Reference

SUMMARY:
This study is a randomized, open-label, single dose, crossover study to evaluate the pharmacokinetic profiles and safety of CKD-386 in healthy volunteers under fasting conditions.

DETAILED DESCRIPTION:
To 30 healthy subjects, following treatments are administered dosing in each period and wash-out period is a minimum of 14 days Pharmacokinetic blood samples are collected up to 72hrs. The pharmacokinetic characteristics and safety are assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults volunteers aged ≥19 years
2. Individuals who had 18 kg/m2 ≤ Body Mass Index(BMI) < 30 kg/m2 and total body weight ≥ 55 kg BMI = Weight(kg)/ Height(m)2
3. Following vital signs results at screening

   * Systolic blood pressure: 90 mmHg to 139 mmHg
   * Diastolic blood pressure: 60 mmHg to 89 mmHg
4. Individuals without congenital/chronic diseases and without abnormal symptoms or diagnosis based on a medical examination
5. Individuals who were deemed to be appropriate as study subjects following laboratory tests (hematology, blood chemistry, serology, urology etc.) and ECG etc. performed
6. Individuals who agreed proper contraception during the study and did consent to not donation of sperm or eggs 14 days after the last dose of study drug
7. Individuals who signed an informed consent form after being fully informed of the study prior to participation, including the objective and content

Exclusion Criteria:

1. Individuals who had been administered investigational product(s) from other clinical study or bioequivalence study within the 6 months prior to the first administration of investigational drugs
2. Those who have used drugs that induce or inhibit drug metabolizing enzymes, such as barbiturates, within 1 month before the first dosing date, or who have used drugs that may interfere with this study within 10 days before the first dosing day (However, clinical investigational drugs) Participation is possible in consideration of pharmacokinetic and pharmacodynamic characteristics such as interaction with concomitant drugs and half-life of concomitant drugs)
3. Individuals who donated whole blood within the 8 weeks, or blood components within 4 weeks or had a blood transfusion within 4 weeks prior to the first administration of investigational drugs
4. Individuals who have a history of gastrointestinal surgery except simple appendectomy and hernia surgery
5. Individuals who meet the following condition with 1 month of the first administration of investigational drugs

   * Alcohol: Man-21 glasses/week, Woman-14 glasses/week (1 glass = soju 50mL or liquor 30mL or beer 250mL)
   * Smoking: 20 cigarettes/day
6. Patients with the following diseases

   * Patients with hypersensitivity to the main constituents or components of the investigational drug
   * Severe hepatic impairment, biliary atresia or cholestasis
   * Patients with hereditary angioedema or with a history of angioedema in the treatment of ACE inhibitors or angiotensin II receptor antagonists
   * Diabetes mellitus
   * Patients with moderate to severe renal impairment [glomerular filtration rate (eGFR) <60 mL / min / 1.73m^2]
   * Renal vascular hypertension patients
   * Patients with active liver disease, including unexplained persistent serum transaminase elevations or elevated serum transaminase elevations greater than three times the normal upper limit
   * Patients with myopathy or have a history of family or genetic history of myopathy
   * Hypothyroidism
   * If you have a history of muscle toxicity for other HMG-CoA converting enzymes or fibrate class drugs
7. Individuals who have genetic problems such as galactose intolerance, Lap lactase deficiency, or glucose-galactose malabsorption
8. Those who are deemed insufficient to participate in this clinical study by investigators
9. Woman who are pregnant or breastfeeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2022-09-23 (Actual); Primary Completion 2022-11-27 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
AUCt of CKD-386 | 0, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72 hours
  Area under the CKD-386 concentration in blood-time curve from 0 to t
Cmax of CKD-386 | 0, 0.25, 0.5, 0.75, 1, 1.25, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 48, 72 hours
  The maximum CKD-386 concentration in blood sampling time t

CONTACTS AND LOCATIONS:
Overall Officials: Jaewoo Kim, M.D., Principal Investigator — Gwanak-gu, Seoul, South Korea, 08779
Locations (1):
- H+ Yangji Hospita, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No